CLINICAL TRIAL: NCT01086319
Title: Comparison of Risk of Hospitalization for Severe Hypersensitivity (Including Severe Cutaneous Reactions) Between Patients With Type 2 Diabetes Initiating Saxagliptin and Those Initiating Other Oral Antidiabetic Treatments
Brief Title: Risk of Hospitalization for Severe Hypersensitivity (Including Severe Skin Reactions) in Patients With Type 2 Diabetes Exposed to Oral Antidiabetic Treatments
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CV181-103
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed to saxagliptin
- Patients exposed to oral antidiabetic drugs (not saxagliptin)

SUMMARY:
The purpose of this study is to compare the incidence hospitalization for severe hypersensitivity and cutaneous reactions among patients with type 2 diabetes who are new users of saxagliptin and those who are new users of other oral antidiabetic drugs.

DETAILED DESCRIPTION:
Prospectively designed retrospective database study. This study will be conducted using administrative claims data and electronic medical records that are collected as part of routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly prescribed saxagliptin or an Oral Anti-diabetic Drug (OAD) in a class other than Dipeptidyl peptidase IV (DPP4) inhibitors
* Enrolled in the respective database for at least 180 days prior to first prescription of new OAD
* Have at least one diagnostic code for a type 2 diabetes-related condition

Exclusion Criteria:

* Patients with an inpatient diagnostic code for any of the conditions of interest within the 180-day baseline period
* Patients prescribed a DPP4 inhibitor during the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out using databases containing administrative claims data (HealthCore Integrated Research DatabaseSM (HIRD) and Medicare in the U.S.) and electronic medical records (General Practice Research Database (GPRD) and The Health Improvement Network (THIN) in the UK). The US population includes patients from health plans in the northeast, southeastern, mid-Atlantic, central, mid-western, and western regions (HIRD) as well as US citizens 65 years of age and older (Medicare). The UK population includes patients seeking medical care from general practitioners (GPRD and THIN)
Sampling Method: Non-Probability Sample
Enrollment: 113505 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hospitalizations with any hypersensitivity reaction, including anaphylaxis, angioedema, generalized urticaria, SJS, TEN, and other severe skin reactions (i.e., acute generalized exanthematous pustulosis and drug rash with eosinophilia/systemic symptoms) | 12-months
Hospitalizations with any hypersensitivity reaction, including anaphylaxis, angioedema, generalized urticaria, SJS, TEN, and other severe skin reactions (i.e., acute generalized exanthematous pustulosis and drug rash with eosinophilia/systemic symptoms) | 18-months
Hospitalizations with any hypersensitivity reaction, including anaphylaxis, angioedema, generalized urticaria, SJS, TEN, and other severe skin reactions (i.e., acute generalized exanthematous pustulosis and drug rash with eosinophilia/systemic symptoms) | 36-months
Hospitalizations with any hypersensitivity reaction, including anaphylaxis, angioedema, generalized urticaria, SJS, TEN, and other severe skin reactions (i.e., acute generalized exanthematous pustulosis and drug rash with eosinophilia/systemic symptoms) | 54-months

SECONDARY OUTCOMES:
Hospitalized for anaphylaxis | 12-months
Hospitalized for anaphylaxis | 18-months
Hospitalized for anaphylaxis | 36-months
Hospitalized for anaphylaxis | 54-months
Hospitalized for angioedema | 12-months
Hospitalized for angioedema | 18-months
Hospitalized for angioedema | 36-months
Hospitalized for angioedema | 54-months
Hospitalized for generalized urticaria | 12-months
Hospitalized for generalized urticaria | 18-months
Hospitalized for generalized urticaria | 36-months
Hospitalized for generalized urticaria | 54-months
Hospitalized for severe skin reactions | 12-months
Hospitalized for severe skin reactions | 18-months
Hospitalized for severe skin reactions | 36-months
Hospitalized for severe skin reactions | 54-months
Hospitalized for all endpoints | 12-months
Hospitalized for all endpoints | 18-months
Hospitalized for all endpoints | 36-months
Hospitalized for all endpoints | 54-months
Hospitalized/emergency room (ER) visits for hypersensitivity reactions | 12-months
Hospitalized/emergency room (ER) visits for hypersensitivity reactions | 18-months
Hospitalized/emergency room (ER) visits for hypersensitivity reactions | 36-months
Hospitalized/emergency room (ER) visits for hypersensitivity reactions | 54-months
Death from hypersensitivity reactions | 12-months
Death from hypersensitivity reactions | 18-months
Death from hypersensitivity reactions | 36-months
Death from hypersensitivity reactions | 54-months
Hospitalized for Stevens-Johnson syndrome (SJS) | 12-months
Hospitalized for Stevens-Johnson syndrome (SJS) | 18-months
Hospitalized for Stevens-Johnson syndrome (SJS) | 36-months
Hospitalized for Stevens-Johnson syndrome (SJS) | 54-months
Hospitalized for for toxic epidermal necrolysis (TEN) | 12-months
Hospitalized for for toxic epidermal necrolysis (TEN) | 18-months
Hospitalized for for toxic epidermal necrolysis (TEN) | 36-months
Hospitalized for for toxic epidermal necrolysis (TEN) | 54-months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Lo Re V, Carbonari DM, Saine ME, Newcomb CW, Roy JA, Liu Q, Wu Q, Cardillo S, Haynes K, Kimmel SE, Reese PP, Margolis DJ, Apter AJ, Reddy KR, Hennessy S, Bhullar H, Gallagher AM, Esposito DB, Strom BL. Postauthorization safety study of the DPP-4 inhibitor saxagliptin: a large-scale multinational family of cohort studies of five outcomes. BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000400. doi: 10.1136/bmjdrc-2017-000400. eCollection 2017. PMID 28878934
- [Derived] Saine ME, Carbonari DM, Newcomb CW, Nezamzadeh MS, Haynes K, Roy JA, Cardillo S, Hennessy S, Holick CN, Esposito DB, Gallagher AM, Bhullar H, Strom BL, Lo Re V 3rd. Determinants of saxagliptin use among patients with type 2 diabetes mellitus treated with oral anti-diabetic drugs. BMC Pharmacol Toxicol. 2015 Apr 2;16:8. doi: 10.1186/s40360-015-0007-z. PMID 25889498
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4449&filename=CV181_103.pdf